CLINICAL TRIAL: NCT02161133
Title: Cognitive Rehabilitation for Gulf War Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPLD-009-13S
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Gulf War Illness
Keywords: Veterans; neuropsychology; fatigue; Chronic Multisymptom Illness; Gulf War Illness; behavioral treatment
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Problem-Solving Therapy (Experimental): Problem-Solving Therapy is a treatment approach that teaches patients strategies to address real-life problems.
  Interventions: Behavioral: Problem-Solving Therapy
- Health Education (Active Comparator): Health education provides didactic information about Gulf War Illness
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Problem-Solving Therapy — Problem-Solving Therapy is a treatment approach that teaches patients strategies to address real-life problems.
  Arms: Problem-Solving Therapy
Behavioral: Health Education — Health Education provides didactic information about Gulf War Illness
  Arms: Health Education

SUMMARY:
There are almost 700,000 Gulf War Veterans (GWV) with 25-30% suffering from a devastating multi-symptom illness coined Gulf War Illness (GWI). GWV with GWI report significant activity limitations and chronic cognitive problems consistent with problem-solving deficits. Problem-solving is considered the most complex of cognitive abilities and is what enables us to conduct complicated behaviors such as setting goals, sequencing and multi-tasking. As a result studies have found that problem-solving deficits are prospectively related to a greater risk of disability. Despite published reports documenting these problems there are no treatments that target the problem-solving deficits of GWI. This proposal seeks to determine whether Problem-Solving Therapy, a patient centered cognitive rehabilitation therapy, can reduce disability by compensating for problem-solving deficits.

DETAILED DESCRIPTION:
Gulf War Illness (GWI) is a complex multi-dimensional illness which causes as much disability as other major medical diseases. Previous clinical trials (i.e. cognitive behavioral therapy and graded exercise) for GWI have sought to improve disability by increasing activity regardless of symptom presentation. These previous trials for GWI have shown limited efficacy and poor adherence. An innovative treatment approach is to target a specific component of GWI, namely problem-solving ability, known to be associated with disability.

Impairment in problem-solving ability affects Gulf War Veterans (GWV) with GWI and is prospectively related to greater risk of disability. This impairment is also related to poorer adherence to medical regimes, making it difficult for GWV to manage other aspects of GWI. Problem-solving is considered one of the most complex of cognitive abilities and is related to complicated behaviors such as setting goals, sequencing and multi-tasking. Despite published reports documenting these deficits there are no treatments that target the problem-solving deficits of GWI in order to reduce disability.

The investigators propose a targeted treatment, Problem-Solving Therapy, to compensate for the problem-solving deficits of GWI and thereby reducing disability. Problem-Solving Therapy, a top down approach, teaches patients skills to overcome problems like cognitive dysfunction or physical symptoms that impact problem-solving. Compensating for problem-solving deficits would reduce disability and provide information on the effect of treating one component of GWI on other symptoms of GWI. This is the first trial of cognitive rehabilitation therapy for GWI.

ELIGIBILITY:
Inclusion Criteria:

Inclusion:

* deployed to first Gulf War and meets Kansas definition for GWI (see definition in measures section);
* scores at least a half a standard deviation worse than the mean on the World Health Organization Disability Schedule (WHO-DAS II).

Exclusion Criteria:

Exclusion:

* current suicidal/homicide intent or plan assessed by The Columbia Suicide Severity Rating Scale, schizophrenia or current psychotic symptoms
* self-reported diagnosis of a degenerative brain disorder or serious psychiatric or medical illness which may limit generalizability of the findings, limit safety or account for the symptoms of GWI.

Exclusionary medical illnesses include: Class 3 and 4 heart failure, cancer diagnosed within the past year and/or undergoing active treatment (chemotherapy or radiation therapy), chronic renal insufficiency, hospitalization due to myocardial infarct, stroke in the past year, a neurodegenerative disorder, or another medical or psychiatric disorder that may limit generalizability, limit participants safety or account for the symptoms of GWI at the discretion of the PI.

* a disability that would preclude telephone use.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M McAndrew, PhD, Principal Investigator — East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ
Locations (3):
- United States (3):
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey
  - Canandaigua VA Medical Center, Canandaigua, NY, Canandaigua, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sullivan N, Schorpp H, Crosky S, Thien S, Helmer DA, Litke DR, Pigeon WR, Quigley KS, McAndrew LM. Treatment and life goals among veterans with Gulf War illness. PLoS One. 2023 Nov 30;18(11):e0295168. doi: 10.1371/journal.pone.0295168. eCollection 2023. PMID 38033143
- [Derived] Kane NS, Hassabelnaby R, Sullivan NL, Graff F, Litke DR, Quigley KS, Pigeon WR, Rath JF, Helmer DA, McAndrew LM. Veteran Beliefs About the Causes of Gulf War Illness and Expectations for Improvement. Int J Behav Med. 2024 Feb;31(1):169-174. doi: 10.1007/s12529-023-10166-1. Epub 2023 Mar 27. PMID 36973578
- [Derived] Winograd DM, Hyde JK, Bloeser K, Santos SL, Anastasides N, Petrakis BA, Pigeon WR, Litke DR, Helmer DA, McAndrew LM. Exploring the acceptability of behavioral interventions for veterans with persistent "medically unexplained" physical symptoms. J Psychosom Res. 2023 Apr;167:111193. doi: 10.1016/j.jpsychores.2023.111193. Epub 2023 Feb 14. PMID 36822031
- [Derived] McAndrew LM, Quigley KS, Lu SE, Litke D, Rath JF, Lange G, Santos SL, Anastasides N, Petrakis BA, Greenberg L, Helmer DA, Pigeon WR. Effect of Problem-solving Treatment on Self-reported Disability Among Veterans With Gulf War Illness: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2245272. doi: 10.1001/jamanetworkopen.2022.45272. PMID 36472870
- [Derived] Sullivan N, Phillips LA, Pigeon WR, Quigley KS, Graff F, Litke DR, Helmer DA, Rath JF, McAndrew LM. Coping with Medically Unexplained Physical Symptoms: the Role of Illness Beliefs and Behaviors. Int J Behav Med. 2019 Dec;26(6):665-672. doi: 10.1007/s12529-019-09817-z. PMID 31701389

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Problem-Solving Therapy | Health Education
Started | 135 | 133
Completed | 116 | 122
Not Completed | 19 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Problem-Solving Therapy | Health Education | Total
Number analyzed (Participants) | 135 | 133 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (7.6) | 52.8 (7.0) | 52.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 120 | 117 | 237
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 118 | 115 | 233
  Unknown or Not Reported | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 12
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 30 | 33 | 63
  White | 91 | 88 | 179
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 135 | 133 | 268
World Health Organization DIsability Assessment Schedule 2.0 [Mean (Standard Deviation); unit: units on a scale] — World Health Organization Disability Assessment Schedule.
  The WHO-DAS 2.0 measures disability due to physical and mental health conditions. It reflects two underlying constructs: Activity limitations and Participation deficits. Scores range from 0-100 with higher scores = more disability.
  units on a scale | 46 (18.1) | 44.8 (19.1) | 45.4 (18.6)

OUTCOME MEASURES:

1. Primary Outcome: Disability - WHO-DAS 2 Change
Description: World Health Organization Disability Assessment Schedule.
  The WHO-DAS 2.0 measures disability due to physical and mental health conditions. The WHO-DAS 2.0 is a 36 item measure that focuses upon six life tasks:
  * Understanding and communicating
  * Self-care
  * Mobility (getting around)
  * Interpersonal relationships (getting along with others)
  * Work and household roles (life activities)
  * Community and civic roles (participation)
  These six life tasks reflect two underlying constructs: Activity limitations and Participation deficits. Scores range from 0-100 with higher scores = more disability.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Problem-Solving Therapy | Health Education
Number analyzed (Participants) | 116 | 122
score on a scale | -2.81 (1.16) | -2.21 (1.12)
Statistical Analysis 1: Comparison: Problem-Solving Therapy vs Health Education; Test type: Superiority; p = 0.712, Mixed Models Analysis; Mean Difference (Final Values) = -0.60, Standard Error of Mean 1.62

2. Secondary Outcome: Problem-Solving Inventory Change
Description: Self-report problem-solving ability. Scores range from 32-192 with lower scores equally better problem-solving ability.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Problem-Solving Therapy | Health Education
Number analyzed (Participants) | 116 | 122
score on a scale | -12.77 (1.77) | -6.53 (1.74)
Statistical Analysis 1: Comparison: Problem-Solving Therapy vs Health Education; Test type: Superiority; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = -6.18, Standard Error of Mean 2.48

3. Secondary Outcome: Problem-Solving Ability Change
Description: Neuropsychological Battery includes: Halstead Category Test, Russell Revised Version, The Conner's Continuous Performance Test-3 (CPT-3), Stroop Color and Word Test, Trails Making Test A and B (TMT). Problem-solving ability was be created by standardizing (i.e., converting to z-scores) these neuropsychological tests based on administrative norms and averaging them. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population and higher scores reflecting greater problem solving.
Time Frame: Baseline and 12 weeks
Population: Participants who were unable to come in person did not complete this measure, as a result the overall number analyzed was smaller.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Problem-Solving Therapy | Health Education
Number analyzed (Participants) | 75 | 86
score on a scale | 13.81 (7.5) | 1.58 (7.29)
Statistical Analysis 1: Comparison: Problem-Solving Therapy vs Health Education; Test type: Superiority; p = 0.244, Mixed Models Analysis; Mean Difference (Final Values) = 12.23, Standard Error of Mean 10.45

4. Secondary Outcome: Disability - WHO-DAS 2 Change
Description: as for outcome 1
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Problem-Solving Therapy | Health Education
Number analyzed (Participants) | 116 | 122
score on a scale | -2.61 (1.45) | 1.11 (1.29)
Statistical Analysis 1: Comparison: Problem-Solving Therapy vs Health Education; Test type: Superiority; p = 0.057, Mixed Models Analysis; Mean Difference (Final Values) = -3.71, Standard Error of Mean 1.95

5. Other Pre Specified Outcome: Pain Disability Change
Description: Pain Disability Index (PDI). Scale ranges from 0-70 with higher scores meaning worse disability.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Problem-Solving Therapy | Health Education
Number analyzed (Participants) | 116 | 122
score on a scale | -2.05 (1.13) | -0.68 (1.09)
Statistical Analysis 1: Comparison: Problem-Solving Therapy vs Health Education; Test type: Superiority; p = 0.382, Mixed Models Analysis; Mean Difference (Final Values) = -1.37, Standard Error of Mean 1.57

6. Other Pre Specified Outcome: Multidimensional Pain Inventory - Pain Severity Subscale Change
Description: three items assessing pain severity. scores range 0-18 with higher scores=worse severity
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Problem-Solving Therapy | Health Education
Number analyzed (Participants) | 116 | 122
score on a scale | 0 (0.10) | -0.06 (0.10)
Statistical Analysis 1: Comparison: Problem-Solving Therapy vs Health Education; Test type: Superiority; p = 0.703, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, Standard Error of Mean 0.14

7. Other Pre Specified Outcome: Fatigue Change
Description: The Fatigue Severity Scale (FSS). Scale from 9 to 63 with higher scores = worse fatigue
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Problem-Solving Therapy | Health Education
Number analyzed (Participants) | 116 | 122
score on a scale | -2.71 (0.98) | -0.82 (0.95)
Statistical Analysis 1: Comparison: Problem-Solving Therapy vs Health Education; Test type: Superiority; p = 0.168, Mixed Models Analysis; Mean Difference (Final Values) = -1.88, Standard Error of Mean 1.36

8. Secondary Outcome: Problem-Solving Inventory Change
Description: Self-report problem-solving ability. Scores range from 32-192 with lower scores equally better problem-solving ability.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Problem-Solving Therapy | Health Education
Number analyzed (Participants) | 116 | 122
score on a scale | -7.03 (2.91) | 0.26 (1.94)
Statistical Analysis 1: Comparison: Problem-Solving Therapy vs Health Education; Test type: Superiority; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = -7.28, Standard Error of Mean 2.93

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Problem-Solving Therapy | Health Education
All-Cause Mortality (participants affected / at risk) | 1/135 | 0/133
Serious Adverse Events (participants affected / at risk) | 21/135 | 31/133
Other Adverse Events (participants affected / at risk) | 15/135 | 14/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Problem-Solving Therapy (N=135) | Health Education (N=133)
increasing emotionally labile, tearful, disorganized thinking (Psychiatric disorders) | 0 (0) | 1 (1)
increased nightmares (Psychiatric disorders) | 0 (0) | 1 (1)
ER visit (Gastrointestinal disorders) | 1 (1) | 1 (2)
ER Visit (General disorders) | 4 (4) | 4 (4)
Admitted to hospital for numbness in arm (Nervous system disorders) | 1 (1) | 0 (0)
Admitted to hospital for severe abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Admitted to hospital for pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Scheduled plastic surgery (General disorders) | 0 (0) | 1 (1)
ER Visit (Nervous system disorders) | 0 (0) | 2 (2)
ER Visit (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Kidney removed; no chemo or radiation at this time (Surgical and medical procedures) | 0 (0) | 1 (1)
Unplanned surgery for intestinal blockage. (Surgical and medical procedures) | 0 (0) | 1 (1)
Overwhelmed from reflecting about GWI Sx. Felt better after journaling. (Psychiatric disorders) | 0 (0) | 1 (1)
Emotional difficulty during QI. Nighmares after Baseline Visit. (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalized for abdominal pain; Dx with hernia and discharged 3 days after (General disorders) | 1 (1) | 0 (0)
Admitted to hospital for passing out on motorcycle. (General disorders) | 0 (0) | 1 (1)
Hospitalized for same day posterior cervical laminectomy surgery. (Surgical and medical procedures) | 0 (0) | 1 (1)
Increased depression and Suicidal Ideation. Has chronic SI. (Psychiatric disorders) | 1 (1) | 0 (0)
Cataract surgery; overnight stay. Increased dizziness. (Eye disorders) | 1 (1) | 0 (0)
Hospital same day surgery for cyst removal from lower back. (Surgical and medical procedures) | 0 (0) | 1 (1)
Increase in intensity of suicidal ideation without intent. Has a history of SI. (Psychiatric disorders) | 0 (0) | 1 (1)
Increased headaches; previous unreported passive SI when experience headache episode. (Psychiatric disorders) | 1 (1) | 0 (0)
ER Visit (Psychiatric disorders) | 0 (0) | 2 (2)
Hysterectomy surgery and overnight stay at hospital. ER on different day for abnormal amount of blee (Surgical and medical procedures) | 0 (0) | 1 (1)
Dx with Kidney cancer; operation to remove cancer - hospitalized 2 days. (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip replacement and diagnosed with heart disease approx. 1 month after hip replacement (General disorders) | 1 (1) | 0 (0)
Right nephrectomy due to mass found in kidney. Hospitalized for 2 days and discharged. (Surgical and medical procedures) | 1 (1) | 0 (0)
Increased suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
ER Visit (Cardiac disorders) | 0 (0) | 6 (6)
ER Visit (Social circumstances) | 6 (6) | 0 (0)
ER Visit (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Problem-Solving Therapy (N=135) | Health Education (N=133)
distressing memories (Psychiatric disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Chest spasms (Cardiac disorders) | 0 (0) | 1 (1)
Foot issue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hand numbness (Nervous system disorders) | 1 (1) | 0 (0)
Sinusitis/bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Herniated disk (General disorders) | 0 (0) | 1 (1)
Extreme pain and heat in body (General disorders) | 0 (0) | 1 (1)
Heartburn, vertigo (General disorders) | 1 (1) | 0 (0)
Excessive daytime sleepiness (General disorders) | 1 (1) | 0 (0)
Cramping L hand and R foot (General disorders) | 1 (1) | 0 (0)
Rash on face, affecting eyes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Left shoulder pain (Nervous system disorders) | 0 (0) | 1 (1)
Rash on left ear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mononucleosis (Social circumstances) | 0 (0) | 1 (1)
Recurrence of IBS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain up R arm and hand (Nervous system disorders) | 1 (1) | 0 (0)
Increased frequency of nightmares as a result of increasing social activities (Psychiatric disorders) | 1 (1) | 0 (0)
Trouble with memory - signing name (Nervous system disorders) | 0 (0) | 1 (1)
Torn bicep muscle playing ball (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thrown out back from building shelves and drawers. (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Increased pain and sciatica due to increased exercise on treadmill/stationary bike. (Nervous system disorders) | 0 (0) | 1 (1)
Increasing arthritis pain in foot since car accident 3 months ago. (Nervous system disorders) | 1 (1) | 0 (0)
ER Visit (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased frequency of nightmares to 1/week from 3-4 times/year. (Psychiatric disorders) | 0 (0) | 1 (1)
Passive SI without intent or plan. (Psychiatric disorders) | 1 (1) | 0 (0)
PTSD symptoms (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT02161133/Prot_SAP_000.pdf